CLINICAL TRIAL: NCT02706587
Title: Neuromuscular Electrical Stimulation for Intensive Care Unit-acquired Weakness
Brief Title: Neuromuscular Electrical Stimulation for Intensive Care Unit-acquired Weakness Assessment
Acronym: ENS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Fondation Paul Bennetot (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REA 01-2014
Record Dates: First submitted 2016-02-10; First posted 2016-03-11 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Polyneuropathy, Critical Illness
Keywords: Critical illness polyneuropathy; Neuromuscular Electrical Stimulation
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular electrical stimulation (Experimental): NEMS is delivered bilaterally to the quadriceps femoris muscle using a portable battery-powered stimulator (Rehab 400, Cefar Compex, France). The electrodes are placed on the motor points of vastus medialis and vastus lateralis muscles. Electrical stimuli of 45Hz (pulse width: 380 µseconds; 6 seconds on with 1.5 second rise time; and 0.75 seconds fall time.; 5 seconds off). The current is adjusted to ensure maximum tolerable muscle contraction The protocol is applied twice daily for 25 minutes, five days a week.
  Interventions: Device: Neuromuscular electrical stimulation
- Sham Control (Sham Comparator): No electrostimulation
  Interventions: Device: Sham control

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — NEMS is delivered bilaterally to the quadriceps femoris muscle using a portable battery-powered stimulator (Rehab 400, Cefar Compex, France). The electrodes are placed on the motor points of vastus medialis and vastus lateralis muscles. Electrical stimuli of 45Hz (pulse width: 380 µseconds; 6 seconds on with 1.5 second rise time; and 0.75 seconds fall time.; 5 seconds off). The current is adjusted to ensure maximum tolerable muscle contraction The protocol is applied twice daily for 25 minutes, five days a week.
  Arms: Neuromuscular electrical stimulation
Device: Sham control — No electrostimulation
  Arms: Sham Control

SUMMARY:
The purpose of this study is to determine whether early neuromuscular electrical stimulation is effective in the prevention of neuromuscular weakness in critical ill patients.

DETAILED DESCRIPTION:
Randomized, controlled study of early electrical neurostimulation (vs sham) in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All patient
* Aged of 18 or more
* With an intended ICU stay of at least 72 hours
* Mechanically ventilated

Exclusion Criteria:

* Age less than 18 years
* Pregnant women
* Preexisting neuromuscular disease
* Patient bearing a pace maker or an implantable defibrillator.
* Poly traumatism and/or leg fracture.
* End stage disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Medical resuscitation council (MRC) score | up to 25 months. From date of randomization to the date of ICU discharge

SECONDARY OUTCOMES:
Total duration of mechanical ventilation (days) | up to 25 months. From date of randomization to the date of ICU discharge
Length of ICU stay and hospital stay. | up to 25 months. From date of randomization to the date of ICU discharge or hospital discharge
Type of hospital discharge | up to 25 months. From date of randomization to the date of hospital discharge
  (alive/deceased/rehabilitation/home...)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lamer, MD, Principal Investigator — Institut Mutualiste Montsouris, Paris, France
Locations (1):
- Insitut Mutualiste Montsouris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Routsi C, Gerovasili V, Vasileiadis I, Karatzanos E, Pitsolis T, Tripodaki E, Markaki V, Zervakis D, Nanas S. Electrical muscle stimulation prevents critical illness polyneuromyopathy: a randomized parallel intervention trial. Crit Care. 2010;14(2):R74. doi: 10.1186/cc8987. Epub 2010 Apr 28. PMID 20426834
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Needham DM, Truong AD, Fan E. Technology to enhance physical rehabilitation of critically ill patients. Crit Care Med. 2009 Oct;37(10 Suppl):S436-41. doi: 10.1097/CCM.0b013e3181b6fa29. PMID 20046132
- [Background] Kho ME, Truong AD, Brower RG, Palmer JB, Fan E, Zanni JM, Ciesla ND, Feldman DR, Korupolu R, Needham DM. Neuromuscular electrical stimulation for intensive care unit-acquired weakness: protocol and methodological implications for a randomized, sham-controlled, phase II trial. Phys Ther. 2012 Dec;92(12):1564-79. doi: 10.2522/ptj.20110437. Epub 2012 Mar 15. PMID 22421734